CLINICAL TRIAL: NCT01290445
Title: Varenicline Pregnancy Cohort Study Protocol Chantix(Registered)/Champix(Registered) (Varenicline Tartrate)
Brief Title: Varenicline Pregnancy Cohort Study
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: University of Aarhus (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: A3051078
Record Dates: First submitted 2011-01-25; First posted 2011-02-07 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2018-08

CONDITIONS: Malformations
Keywords: varenicline; smoking; smoking cessation; cohort study; drug safety; prospective study
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exposed: Infants exposed in utero to varenicline
  Interventions: Drug: varenicline
- Unexposed: infants exposed in utero to cigarette smoke from maternal smoking
  Interventions: Behavioral: cigarette smoke from maternal smoking
- Reference: infants not exposed in utero to either varenicline or cigarette smoke from maternal smoking
  Interventions: Other: Non-Exposure

INTERVENTIONS:
Drug: varenicline — This is a non-interventional study. Exposure in utero to varenicline is observed, not assigned.
  Other Names: Chantix, Champix
  Groups: Exposed
Behavioral: cigarette smoke from maternal smoking — This is a non-interventional study. Exposure in utero to cigarette smoke from maternal smoking is observed, not assigned.
  Groups: Unexposed
Other: Non-Exposure — This is a non-interventional study. Non-exposure in utero to varenicline and cigarette smoke from maternal smoking is observed, not assigned.
  Groups: Reference

SUMMARY:
A prospective population-based cohort study to examine whether varenicline use during pregnancy is associated with an increased risk of major congenital malformations in infants above that associated with smoking during pregnancy.

DETAILED DESCRIPTION:
Sampling will not be employed. The data sources record nearly all (>98.6%) births in Denmark and Sweden.

ELIGIBILITY:
Inclusion Criteria:

All live and stillbirths between May 2007 and December 2012 in Denmark and Sweden.

Exclusion Criteria:

Births less than 22 weeks of gestation in Denmark and 28 weeks in Sweden are not recorded by the registers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all live born and stillborn infants in Denmark and Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 885185 (Actual)
Dates: Start 2007-09-13 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051078&StudyName=Varenicline%20Pregnancy%20Cohort%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline Exposed Cohort: Participants included infants who were exposed to varenicline in utero.
- Varenicline Unexposed Cohort: Participants included infants who were exposed to maternal smoking, but not to varenicline in utero.
- Reference Cohort: Participants included infants who were neither exposed to maternal smoking nor to varenicline in utero.
Period: Overall Study
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Started | 335 | 78412 | 806438
Completed | 335 | 78412 | 806438
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all infants born in Denmark and Sweden from May 1, 2007 through December 31, 2012.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort | Total
Number analyzed (Participants) | 335 | 78412 | 806438 | 885185
Age, Customized [Number; unit: infants] — Reported age is the gestational age of infants.
  infants
    Less Than (<) 32 weeks | 3 | 1036 | 6275 | 7314
    32-36 weeks | 22 | 5137 | 40457 | 45616
    Greater Than or Equal to (>=) 37 weeks | 310 | 72239 | 759706 | 832255
Sex/Gender, Customized [Number; unit: infants]
  Female | 156 | 38044 | 392755 | 430955
  Male | 179 | 40328 | 413485 | 453992
  Unknown | 0 | 40 | 198 | 238

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants With Major Congenital Malformations
Description: Major congenital malformations were defined as any codes within the Q-chapter of The Tenth Revision of the International Classification of Diseases (ICD-10), excluding certain minor anomalies.
Time Frame: For 12 months after birth
Population: Analysis population included all live born infants in Denmark and Sweden from May 1, 2007 through December 31, 2012.
Measure: Number; unit: infants
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Number analyzed (Participants) | 334 | 78028 | 804020
infants | 12 | 3382 | 33950
Statistical Analysis 1: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Crude prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.46 to 1.47]
Statistical Analysis 2: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Adjusted prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.45 to 1.42]

2. Secondary Outcome: Number of Infants With Stillbirths
Description: Stillbirth was defined as death at a gestational age of greater than or equal to (>=) 22 weeks, with the exception that in Sweden prior to 2008 it was defined as death at a gestational age of >=28 weeks.
Time Frame: At the time of birth
Population: Analysis population included all infants born in Denmark and Sweden from May 1, 2007 through December 31, 2012.
Measure: Number; unit: infants
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Number analyzed (Participants) | 335 | 78412 | 806438
infants | 1 | 384 | 2418
Statistical Analysis 1: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Crude prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.09 to 4.34]
Statistical Analysis 2: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Adjusted prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.09 to 4.67]

3. Secondary Outcome: Number of Infants Born Small for Gestational Age (SGA)
Description: An infant was defined as SGA if birth weight was below the 10th percentile of its sex-specific national distribution at the respective gestational week. Data on birth weight and gestational age from the medical birth registries were used to calculate the 10th percentiles for each sex based on all Danish and Swedish births during the study observation period.
Time Frame: At the time of birth
Population: Analysis population included all infants born in Denmark and Sweden from May 1, 2007 through December 31, 2012.
Measure: Number; unit: infants
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Number analyzed (Participants) | 335 | 78412 | 806438
infants | 42 | 13433 | 73135
Statistical Analysis 1: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Crude prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.50 to 0.96]
Statistical Analysis 2: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Adjusted prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.51 to 0.97]

4. Secondary Outcome: Number of Infants Born Preterm
Description: Preterm birth was defined as birth before the gestational age of 37 weeks.
Time Frame: At the time of birth
Population: Analysis population included all infants born in Denmark and Sweden from May 1, 2007 through December 31, 2012.
Measure: Number; unit: infants
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Number analyzed (Participants) | 335 | 78412 | 806438
infants | 25 | 6173 | 46732
Statistical Analysis 1: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Crude prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.63 to 1.42]
Statistical Analysis 2: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Adjusted prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.61 to 1.37]

5. Secondary Outcome: Number of Infants Born To Mothers Diagnosed With Premature Rupture of Membranes
Time Frame: At the time of birth
Population: Analysis population included all infants born in Denmark and Sweden from May 1, 2007 through December 31, 2012.
Measure: Number; unit: infants
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Number analyzed (Participants) | 335 | 78412 | 806438
infants | 12 | 4246 | 30641
Statistical Analysis 1: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Crude prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.37 to 1.16]
Statistical Analysis 2: Comparison: Varenicline Exposed Cohort vs Varenicline Unexposed Cohort; Adjusted prevalence odds ratios were estimated along with 95% confidence intervals using logistic regression models; Test type: Superiority or Other; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.37 to 1.16]

6. Secondary Outcome: Number of Infants Diagnosed With Sudden Infant Death Syndrome (SIDS)
Description: Sudden Infant Death Syndrome (SIDS) was defined as a sudden unexplained death of an infant less than one year of age.
Time Frame: For 12 months after birth
Population: Analysis population included all infants born in Denmark and Sweden from May 1, 2007 through December 31, 2012. Here, 'Number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: infants
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Number analyzed (Participants) | 307 | 71720 | 755939
infants | 0 | 51 | 58

ADVERSE EVENTS:
Description: Since this was a non interventional study using secondary data sources, collection and reporting of adverse events were not applicable.
Arm/Group | Varenicline Exposed Cohort | Varenicline Unexposed Cohort | Reference Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.